CLINICAL TRIAL: NCT06469554
Title: Effect of a Multicomponent Exercise Program With Virtual Reality (MEP-VR) Versus Standard Approaches on Functional and Cognitive Domains in Hospitalised Geriatric Patients: Study Protocol for a Randomized Controlled Trial
Brief Title: Effect of a Multicomponent Exercise Program With Virtual Reality (MEP-VR) vs Standard Approaches on Functional and Cognitive Domains in Hospitalized Geriatric Patients: Study Protocol for a Randomized Controlled Trial.
Acronym: MEP-VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MEP-VR
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Hospital Acquired Condition; Frailty
Keywords: Hospital-associated functional decline; Cognitive stimulation; Physical exercise; Virtual Reality; Multicomponent exercise program
MeSH Terms: conditions — Iatrogenic Disease; Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants or their caregivers/legal guardians will be informed of their random inclusion in one of the three groups, but they will not be aware of the specific group to which they have been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Group (No Intervention): Participants randomly assigned to this group will receive standard hospital care, which may include physical rehabilitation if deemed necessary by the clinical staff.
- Intervention group (Experimental): Participants in this group will receive a Multicomponent Exercise Program (MEP) or with virtual reality added
  Interventions: Behavioral: MEP-only group; Behavioral: MEP-VR group

INTERVENTIONS:
Behavioral: MEP-only group — Participants in this group will receive a Multicomponent Exercise Program (MEP) consisting of: Supervised aerobic training on a stationary bike Progressive resistance/strength training using weight machines Balance training exercises The MEP sessions will be 30-40 minutes long and conducted over 4 consecutive days.
  Arms: Intervention group
Behavioral: MEP-VR group — Participants in this group will receive the same MEP intervention as the MEP-only group.
  Additionally, they will use an immersive virtual reality (IVR) system during the exercise program
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to test the effectiveness of a Multicomponent Exercise Program with Virtual Reality (MEP-VR) compared to a Multicomponent Exercise Program (MEP-only) or usual care, in terms of functional and cognitive outcomes in hospitalized older adults.

The main questions it aims to answer are:

* Does the MEP-VR program improve the functionality of hospitalized older adults compared to the other groups?
* Does the MEP-VR program improve the cognitive, mood, and quality of life outcomes of hospitalized older adults compared to the other groups?

Participants will be randomly assigned to one of three groups: a control group or one of the two intervention groups. The intervention groups will receive either the MEP-VR or MEP-only program, which consists of supervised aerobic exercise, resistance training, and balance training, with or without a virtual reality component designed specifically for this study. The intervention will take place over four consecutive days, with each session lasting 30-40 minutes.

The primary outcome will be the functional changes at the time of discharge. Cognition, mood, quality of life, and VR usability will also be assessed.

Technological advances are rapidly increasing with population aging, creating potential benefits for integrating technology into the care of older adults. This study comprehensively evaluates the implementation of VR combined with the multicomponent exercise program. If the hypothesis is confirmed, it would pave the way for modifying the hospitalization system and reducing the critical healthcare burden resulting from the commonly acquired disability in the older population.

DETAILED DESCRIPTION:
Acute hospitalization often leads to functional impairment and disability in older adults as a side effect. Reduced physiological resources increase the risk of negative consequences like functional and cognitive decline, longer hospital stays, and higher mortality and institutionalization rates. Approximately 30-50% of hospitalized older adults experience functional decline, which increases their risk of worsening function or death in the year after discharge.

Conventional care models tend to overlook the negative effects of hospitalization and fail to leverage the potential benefits of technology. Recent studies have found that physical exercise and early rehabilitation programs can prevent functional and cognitive decline during hospitalization and reduce hospital stay and mortality. While Multicomponent Exercise Programs (MEP) that focus on promoting mobility have shown benefits, adding virtual reality (VR) to MEP (MEP-VR) may provide additional physical and cognitive performance improvements in hospitalized patients.

VR is an emerging tool that can engage older adults in physical and cognitive activities. Immersive VR (IVR) systems like head-mounted displays can transport users into virtual environments to execute activities and stimulate cognitive skills. VR is considered an affordable, novel, and safe tool, but further research is needed on its benefits and limitations for older adults.

The main aim of this study is to investigate the effects of MEP-VR on functional and cognitive outcomes in hospitalized older adults compared to standard care. It will also assess the effects on mood, safety, and usability.

Methods

This will be a three-arm randomized clinical trial with two experimental intervention groups (MEP-only, MEP-VR) and a control group (usual care). It will be conducted in the Acute Geriatric Unit (AGU) at a hospital in Spain.

Eligible patients aged 75+ with a Barthel Index score of at least 60, who can walk and cooperate, have an estimated hospital stay of at least 4 days, and provide informed consent, will be randomly assigned to one of the three groups. Those with severe dementia, terminal illness, or clinical instability will be excluded.

The MEP-only group will receive supervised aerobic, resistance, and balance training over 4 consecutive days. The MEP-VR group will receive the same MEP with the addition of IVR components, including using VR during the bike warm-up and while doing resistance exercises. The control group will receive usual care.

Outcomes will be assessed at baseline, end of intervention, and 3 months post-discharge. The primary outcome is functional changes at discharge, measured by the Short Physical Performance Battery, Timed Up and Go, Barthel Index, handgrip strength, and 1-repetition maximum strength tests. Secondary outcomes include cognition, mood, quality of life, and VR-related measures like usability and cybersickness.

The study will be conducted according to randomization and blinding principles. The researcher assigning groups will be different from the attending geriatrician. Patients/caregivers will be blinded to group allocation. Assessors will be blinded but intervention staff will not. Adverse events and dropouts will be recorded.

The study was approved by the ethics committee and registered at ClinicalTrials.gov.

Intervention Details

The MEP-only intervention will consist of:

7-10 min warm-up on a stationary bike 15-20 min resistance training using weight machines 10 min balance training using light-based exercises

The MEP-VR intervention will include the same MEP components plus:

VR during the bike warm-up, allowing patients to virtually tour different locations VR during resistance exercises, with a virtual rural environment displayed The VR system was developed using Unity, C++, OpenXR, and Low Poly graphics for optimal performance and visual comfort The usual care control group will receive standard hospital care, including physical rehabilitation if needed.

Outcomes

Primary outcome: Changes in functional capabilities during the study period, assessed through:

Short Physical Performance Battery Timed Up and Go test Barthel Index Handgrip strength

1-repetition maximum strength tests

Secondary outcomes:

Changes in cognitive function (Mini-Mental State Exam) Changes in mood (Geriatric Depression Scale, Anxiety Inventory) Quality of life (EuroQol-5D-5L) VR-related outcomes (usability, cybersickness, satisfaction) Adverse events, adherence, and perceived exertion Discussion

This study focuses on developing individualized, multicomponent programs to address and prevent functional decline in hospitalized older adults by incorporating innovative technologies like VR. Advances in technology are increasing concurrently with population aging, presenting opportunities to integrate technology into elder care. However, older adults are often excluded from research, leading to limited knowledge on the potential benefits of these technologies.

This randomized trial comprehensively evaluates the implementation of IVR combined with a multicomponent exercise program. It assesses whether IVR can provide greater motivation and willingness to exercise, leading to greater functional and cognitive improvements, as well as impacts on mood, quality of life, and feasibility.

If the hypothesis is confirmed, this project could pave the way for modifying the hospitalization system to leverage technology and help reduce the critical healthcare burden resulting from hospital-acquired disability in older adults

ELIGIBILITY:
Inclusion Criteria:

* Age 75 years or older
* Barthel Index score of at least 60 points
* Able to walk and cooperate
* Estimated hospital stay of at least 4 days
* Able to provide informed consent

Exclusion Criteria:

* Severe dementia
* Terminal illness
* Clinical instability

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The Short Physical Performance Battery (SPPB) | Measured at baseline, end of 4-day intervention, and 3 months post-discharge.
  The Short Physical Performance Battery (SPPB) is a validated instrument used for detecting frailty and predicting disability, institutionalization, and mortality in older adults. It includes the following three tests: Balance tests: Side-by-side stand Semi-tandem stand Tandem stand Gait speed test: Participants are timed walking 4 meters at their usual pace. Chair stand test: Participants are timed as they rise from a chair and return to a seated position five times without using their arms. The SPPB provides a total score ranging from 0 (worst performance) to 12 (best performance) points by summing the scores from each of the three components. Lower SPPB scores indicate poorer physical function and higher risk of adverse health outcomes. The SPPB is a widely used and reliable measure of physical performance in older adults, making it a suitable primary outcome for assessing the functional changes in this study population of hospitalized older individuals
Timed Up and Go (TUG) | The TUG will be administered at the same three time points as the other primary outcome measures: At the start of the 4-day intervention during acute hospitalization At the end of the 4-day intervention 3 months after hospital discharge during the outpa
  The Timed Up and Go (TUG) test is used to assess dynamic balance and risk of falling in older adults. It measures the time in seconds it takes for an individual to get up from a chair, walk 3 meters, and return to the chair

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | through study completion, an average of 1 year
  Cognitive evaluation
Geriatric Depression Scale (GDS): | through study completion, an average of 1 year
  Specifically designed to assess depression in older adults 15-item questionnaire with a scale ranging from 0 (best) to 15 (worst)
State-Trait Anxiety Inventory (STAI) | through study completion, an average of 1 year
  Assesses both state anxiety (current, transient feelings) and trait anxiety (general, long-term tendency) Contains separate scales for state anxiety and trait anxiety Measures overall anxiety levels, not specifically depression
Self-perceived acceptance, usability, and satisfaction using the System Usability Scale | The SUS will be administered during the 4-day intervention period, while the participants are actively using the VR system as part of the MEP-VR program
  The SUS is a 10-question survey that measures a user's subjective assessment of a system's usability on a scale from 1 (lower) to 5 (higher). This validated scale will be used to assess the participants' perceptions of the acceptability, usability, and satisfaction with the VR components integrated into the MEP-VR intervention.
EuroQol-5D-5L questionnaire | through study completion, an average of 1 year
  It consists of two main components: Descriptive system: Assesses five dimensions of health status: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-point scale from 1 (no problems) to 5 (extreme problems). Visual Analogue Scale (VAS): Allows the participant to rate their overall health on a vertical scale from 0 (worst health state imaginable) to 100 (best health state imaginable). The EQ-5D-5L provides a profile of the respondent's health status across the five dimensions, as well as a single index value for their overall health-related quality of life. Timing: In this study, the EQ-5D-5L will be administered at three time points: At the start of the 4-day intervention during acute hospitalization At the end of the 4-day intervention 3 months after hospital discharge during the outpatient follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
Sharing study data upon reasonable request
  Individual participant data (IPD) collected in this randomized controlled trial will be available for sharing upon reasonable request. This includes basic demographic data as well as results from assessments of functionality, cognition, mood, quality of life, and virtual reality experience.
  Researchers interested in accessing these IPD can contact the research team. Requests will be evaluated, and if approved, data will be shared in a timely manner while maintaining participant confidentiality and privacy.
  This data sharing aims to foster scientific collaboration, enable secondary analyses, and replicate the findings, contributing to the advancement of knowledge in geriatric rehabilitation and emerging technologies.
  Instructions for requesting IPD access will be available at [website/research team contact]. All requests will be fairly and transparently reviewed to ensure compliance with ethical and data protection standards.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Instructions for requesting IPD access will be available starting January 2026 at [research team contact]. IPD and supporting information will be available for 5 years, after which requests will no longer be accepted. All requests will be fairly and transparently reviewed to ensure compliance with ethical and data protection standards.
Access Criteria: Sharing study data upon reasonable request
  Individual participant data (IPD) collected in this randomized controlled trial will be available for sharing upon reasonable request. This includes basic demographic data as well as results from assessments of functionality, cognition, mood, quality of life, and virtual reality experience.
  Researchers and qualified investigators will be able to access the IPD and supporting information. Upon request, they will be granted access to:
  Anonymized individual participant-level data Detailed study protocol Statistical analysis plan Annotated case report forms To access the data, researchers will need to submit a formal request to the research team, outlining the intended use of the data. Requests will be evaluated based on scientific merit, conflicts of interest, and compliance with ethical standards. If approved, researchers will be provided secure access to download the relevant files.
URL: https://www.navarrabiomed.es/es/directorio/martinez-velilla

REFERENCES:
- [Derived] Ferrara MC, Zambom-Ferraresi F, Galbete A, Fernandez-Gonzalez de la Riva M, Izco-Cubero M, Garcia-Baztan A, Capon-Saez A, Dominguez-Mendoza S, Marin-Epelde I, Zambom-Ferraresi F, Martinez-Velilla N. Effect of a Multicomponent Exercise Program with Virtual Reality (MEP-VR) versus standard approaches on functional and cognitive domains in hospitalised geriatric patients: Study protocol for a randomized controlled trial. Rev Esp Geriatr Gerontol. 2025 Jul-Aug;60(4):101646. doi: 10.1016/j.regg.2025.101646. Epub 2025 Mar 13. PMID 40086340